CLINICAL TRIAL: NCT01865487
Title: A Phase I/IIa Double-Blind, Randomized, Placebo-controlled Dose-Finding Study to Evaluate the Safety and Immunogenicity of AERAS-456 in HIV-Negative Adults With and Without Latent Tuberculosis Infection
Brief Title: A Phase I/IIa AERAS-456 in HIV-Negative Adults With & Without Latent Tuberculosis Infection (C-035-456)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-035-456
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Latent Tuberculosis Bacteriology and Histology Unknown; Latent Tuberculosis
Keywords: BCG Vaccinated; HIV Negative
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: A 2 phase study based on LTBI status. Phase 1 is a dose ranging study of a 2 dose regimen at 3 dosage levels and placebo in LTBI negative participants. The second phase evaluated 2 and 3 dose regimens and included + and - LTBI participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 2-Dose Placebo (Placebo Comparator): Placebo QFT Neg and Pos, 2 Doses, days 0,56
  Interventions: Biological: Placebo
- 2-Dose 5/500 H56ug/IC31nmol (Experimental): 5/500 H56ug/IC31nmol QFT Neg and Pos, 2 Doses, days 0,56
  Interventions: Biological: H56ug/IC31nmol
- 2-Dose 15/500 H56ug/IC31nmol (Experimental): 15/500 H56ug/IC31nmol QFT Negative 2 Doses, days 0,56
  Interventions: Biological: H56ug/IC31nmol
- 2-Dose 50/500 H56ug/IC31nmol (Experimental): 50/500 H56ug/IC31nmol QFT Negative 2 Doses, days 0,56
  Interventions: Biological: H56ug/IC31nmol
- 3-Dose, Placebo (Placebo Comparator): Placebo QFT Neg and Pos, 3 doses, days 0, 56, 112
  Interventions: Biological: Placebo
- 3-Dose, 5/500 H56ug/IC31nmol (Experimental): 5/500 H56ug/IC31nmol QFT Neg and Pos, 3 Doses, days 0, 56, 112
  Interventions: Biological: H56ug/IC31nmol

INTERVENTIONS:
Biological: H56ug/IC31nmol — H56:IC31 (designated as AERAS-456 for Aeras-sponsored clinical development) contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c) formulated in the Th1-stimulating IC31 adjuvant.
  Other Names: AERAS-456
  Arms: 2-Dose 15/500 H56ug/IC31nmol; 2-Dose 5/500 H56ug/IC31nmol; 2-Dose 50/500 H56ug/IC31nmol; 3-Dose, 5/500 H56ug/IC31nmol
Biological: Placebo — Sterile buffer consisting of 10mM Tris and 169mM NaCl at pH 7.4
  Arms: 2-Dose Placebo; 3-Dose, Placebo

SUMMARY:
This is a Phase I/IIa, double-blind, randomized, placebo-controlled, dose- and regimen-finding study in healthy adults with and without LTBI, who are BCG-vaccinated, HIV negative, and have no history or evidence of TB disease. The investigational product is AERAS-456 at 3 dose levels: 5, 15, and 50ug of H56 antigen with 500 nmol IC31. The vaccine is administered by IM injection.

DETAILED DESCRIPTION:
This is a Phase I/IIa, double-blind, randomized, placebo-controlled, dose- and regimen-finding study in healthy adults with and without latent Tuberculosis (TB) Infection, who are Bacille Calmette Guerin (BCG)-vaccinated, HIV negative, and have no history or evidence of TB disease. The investigational product is AERAS-456 at 3 dose levels: 5, 15, and 50ug of H56 antigen with 500 nmol IC31. The vaccine is administered by intramuscular (IM) injection. The study will be conducted at two sites in South Africa.

A total of 98 subjects will be enrolled in 2 phases into 4 groups based on Latent TB Infection (LTBI) status. The initial phase will be a dose ranging study of a 2-dose regimen at 3 dosage levels in LTBI(-) subjects, to select a dosage for the second phase. In the second phase, the study will be expanded to evaluate both 2-dose and 3-dose regimens and to include LTBI(+) subjects. In the first phase, 50 LTBI(-) subjects will be enrolled in Group 1 and randomized at a ratio of 3:3:3:1 to receive 2 doses of 5/500, 15/500, or 50/500 of AERAS-456, or placebo given at Study Days 0 and 56 (Table 0 1).

One dose level of AERAS-456 will be selected by the sponsor and SSI for the second phase of the study, based on analysis of unblinded safety and immunogenicity data through 28 days after the second dose in the first phase, in conjunction with safety and immunogenicity data from study C-032-456. The criteria for dose-selection will be specified in a statistical analysis plan to be finalized prior to the unblinded review. The selected dose, in conjunction with the unblinded safety and immunogenicity data, will be submitted to the SMC for review. In the second phase, 48 subjects will be enrolled concurrently into Group 2 (LTBI[-]) and into Groups 3 and 4 (LTBI[+], Table 0 2). In each of Groups 2 and 4, 16 subjects will be randomized at a ratio of 3:1 to receive 3 doses of AERAS-456 or placebo given at Study Days 0, 56, and 112. In Group 3, 16 subjects will be randomized at a ratio of 3:1 to receive 2 doses of AERAS-456 or placebo given at Study Days 0 and 56.

All subjects will stay on the study for 292 days after receiving the first vaccination. The subjects in Groups 1 and 3 will be followed up for 236 days after the second vaccination and subjects in Groups 2 and 4 will be followed up for 180 days after the third vaccination. The sample size for each study cohort was selected because it was judged to be adequate for preliminary safety and immunogenicity evaluations for a Phase I/IIa study rather than for statistical reasons. Given 12 and 15 subjects in individual AERAS-456 dosing groups, the study will have an 80% probability of detecting at least 1 specified event which occurs at a rate of 12.5% and 10.0%, respectively. If no such events are observed among 12 and 15 subjects receiving active study vaccine, an approximation to the upper one-sided 95% confidence bound on the rate of occurrence for that event would be 22% and 18%, respectively.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria prior to Study Day 0 vaccination:

1. Has completed the written informed consent process prior to the start of screening evaluations.
2. Is male or female.
3. Is age 18 through 50 years at the time of randomization.
4. Received BCG vaccination at least 5 years prior to randomization.
5. Females: Ability to avoid pregnancy during the trial: Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must avoid pregnancy with an acceptable method of avoiding pregnancy from 28 days prior to administration of the study vaccine through the end of the study.
6. Has general good health, confirmed by medical history and physical examination at screening.
7. Is able and willing to complete the full follow-up period of 292 days as required by the protocol.
8. Agrees to avoid elective surgery for the full duration of the study.
9. [Groups 1 and 2] Does not have LTBI, determined by a negative QFT at screening or[Groups 3 and 4] Has LTBI, determined by a positive QFT at screening.

Exclusion Criteria:

Subjects must meet none of the following criteria prior to Study Day 0 vaccination:

1. Acute illness at the time of randomization.
2. Oral temperature 37.5 degrees C at the time of randomization.
3. Abnormal laboratory values from blood collected within 21 days prior to Study Day 0 vaccination.
4. Abnormal urinalysis that, in the opinion of the investigator, indicates systemic or local disease.
5. History or evidence of tuberculosis disease, including but not limited to pulmonary tuberculosis, pleural tuberculosis, lymph node tuberculosis or tuberculosis meningitis.
6. Received a TST within 21 days prior to a scheduled study vaccination.
7. Received investigational Mtb vaccine at any time prior to Study Day 0.
8. History or evidence of autoimmune disease.
9. History or laboratory evidence of HIV-1 infection at screening.
10. Positive test for hepatitis B surface antigen or hepatitis C antibody at screening.
11. Used immunosuppressive medication (other than inhaled or topical immunosuppressants) within 21 days prior to Study Day 0.
12. Received immunoglobulin or blood products within 21 days prior to Study Day 0.
13. Received any investigational product within 21 days prior to Study Day 0, or plans to participate in any other study involving administration of investigational product during the study period.
14. Inability to discontinue current chronic prescription medications, except contraceptives, inhaled or topical immunosuppressants, or nutritional supplements, during the study period.
15. Documented history of allergic reaction or hypersensitivity to any component of the study vaccine.
16. All female subjects: currently pregnant or lactating/nursing; or positive serum pregnancy test during screening; or positive urine pregnancy test on the day of any study vaccination.
17. History or evidence of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may compromise the safety of the subject in the study or interfere with the evaluation of the safety or immunogenicity of the vaccine.
18. History of dermatologic disease or skin features that, in the opinion of the investigator, may interfere with the assessment of injection site reactions.
19. History or evidence of any medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dereck Tait, MD, Study Director — Aeras; Angelique Luabeya, MD, Principal Investigator — University of Cape Town South African Tuberculosis Vaccine Initiative
Locations (2):
- South Africa (2):
  - eKhayavac TB Vaccine Trial, Khayelitsha, Cape Town
  - SATVI Project Office, Brewelskloof Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suliman S, Luabeya AKK, Geldenhuys H, Tameris M, Hoff ST, Shi Z, Tait D, Kromann I, Ruhwald M, Rutkowski KT, Shepherd B, Hokey D, Ginsberg AM, Hanekom WA, Andersen P, Scriba TJ, Hatherill M; H56-035 Trial Group. Dose Optimization of H56:IC31 Vaccine for Tuberculosis-Endemic Populations. A Double-Blind, Placebo-controlled, Dose-Selection Trial. Am J Respir Crit Care Med. 2019 Jan 15;199(2):220-231. doi: 10.1164/rccm.201802-0366OC. PMID 30092143

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 2-dose 5/500: 5/500 H56ug/IC31nmol, QFT Negative, 2 doses, days 0 and 56
- Group 1: 2-dose 15/500: 15/500 H56ug/IC31nmol, QFT Negative, 2 doses, days 0 and 56
- Group 1: 2-dose 50/500: 50/500 H56ug/IC31nmol, QFT Negative, 2 doses, days 0 and 56
- Group 1: 2-dose Placebo: Placebo, QFT Negative, 2 doses, days 0 and 56
- Group 2: 3-dose 5/500: 5/500 H56ug/IC31nmol, QFT Negative, 3 doses, days 0, 56, 112
- Group 2: 3-dose Placebo: Placebo, QFT Negative, 3 doses, days 0, 56, 112
- Group 3: 2-dose 5/500: 5/500 H56ug/IC31nmol, QFT Positive, 2 doses, Days 0 and 56
- Group 3: 2-dose Placebo: Placebo, QFT Positive, 2 doses, Days 0 and 56
- Group 4: 3-dose 5/500: 5/500 H56ug/IC31nmol, QFT Positive, 3 doses, days 0, 56, 112
- Group 4: 3-dose Placebo: Placebo, QFT positive, 3 doses, Days 0, 56, 112
Period: Overall Study
Arm/Group | Group 1: 2-dose 5/500 | Group 1: 2-dose 15/500 | Group 1: 2-dose 50/500 | Group 1: 2-dose Placebo | Group 2: 3-dose 5/500 | Group 2: 3-dose Placebo | Group 3: 2-dose 5/500 | Group 3: 2-dose Placebo | Group 4: 3-dose 5/500 | Group 4: 3-dose Placebo
Started | 15 | 15 | 15 | 5 | 12 | 4 | 12 | 4 | 12 | 4
Completed | 15 | 15 | 15 | 4 | 11 | 4 | 11 | 4 | 12 | 4
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2-Dose Placebo: Placebo, QFT Neg and Pos, 2 doses day 0 and 56
- 2-Dose 5/500 H56/IC31nmol: 5/500 H56ug/IC31nmol, QFT Neg and Pos, 2 Doses, days 0 and 56
- 2-Dose 15/500 H56/IC31nmol: 15/500 H56ug/IC31nmol, QFT Negative, 2 Doses, days 0 and 56
- 2-Dose 50/500 H56/IC31nmol: 50/500 H56ug/IC31nmol, QFT Negative, 2 Doses, days 0 and 56
- 3-Dose Placebo: Placebo QFT Neg and Pos, 3 Doses, days 0, 56, 112
- 3-Dose 5/500 H56/IC31nmol: 5/500 H56ug/IC31nmol, QFT Neg and Pos, 3 Doses, days 0, 56, 112
- Total: Total of all reporting groups
Arm/Group | 2-Dose Placebo | 2-Dose 5/500 H56/IC31nmol | 2-Dose 15/500 H56/IC31nmol | 2-Dose 50/500 H56/IC31nmol | 3-Dose Placebo | 3-Dose 5/500 H56/IC31nmol | Total
Number analyzed (Participants) | 9 | 27 | 15 | 15 | 8 | 24 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (9.51) | 27.2 (8.71) | 24.3 (4.08) | 25.3 (8.76) | 24.9 (8.25) | 28.4 (8.34) | 26.6 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 19 | 6 | 11 | 6 | 17 | 66
  Male | 2 | 8 | 9 | 4 | 2 | 7 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 6 | 7 | 3 | 8 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coloured | 4 | 18 | 9 | 8 | 5 | 16 | 60
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] — Baseline Body Mass Index in kg/m^2
  kg/m^2 | 26.83 (8.385) | 27.11 (6.655) | 25.74 (8.122) | 31.14 (10.922) | 27.75 (12.612) | 25.56 (5.726) | 27.17 (8.191)
LTBI Status at Baseline [Count of Participants; unit: Participants] — LTBI = Latent tuberculosis infection
  Participants
    LTBI Negative | 5 | 15 | 15 | 15 | 4 | 12 | 66
    LTBI Positivie | 4 | 12 | 0 | 0 | 4 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Unsolicited and Solicited Adverse Events Recorded Post Day 0 Vaccination.
Description: Evaluation of unsolicited and solicited AEs was performed through 28 days after each study vaccination. Serious AEs were collected throughout the entire study period (i.e., 292 days). Evaluation of the safety profile of AERAS-456 was performed using data from all subjects who received at least one dose.
Time Frame: Up to 10 months
Population: Safety analysis set
Measure: Number; unit: Participants
Groups:
- Placebo QFT Neg: 2-doses and 3-doses (Groups 1 and 2)
- Placebo QFT Pos: 2-doses and 3-doses (Groups 3 and 4)
- 2-Doses 5/500 QFT Neg; 2-Doses 15/500; 2-Doses 50/500: QFT Negative (Group 1)
- 3-Doses 5/500 QFT Neg: QFT Negative (Group 2)
- 2-Doses 5/500 QFT Pos: QFT Positive (Group 3)
- 3-Doses 5/500 QFT Pos: QFT Positive (Group 4)
Arm/Group | Placebo QFT Neg | Placebo QFT Pos | 2-Doses 5/500 QFT Neg | 2-Doses 15/500 | 2-Doses 50/500 | 3-Doses 5/500 QFT Neg | 2-Doses 5/500 QFT Pos | 3-Doses 5/500 QFT Pos
Number analyzed (Participants) | 9 | 8 | 15 | 15 | 15 | 12 | 12 | 12
Participants
  Participants with AEs | 7 | 8 | 15 | 15 | 15 | 10 | 10 | 10
  Participants with related AEs | 5 | 4 | 12 | 11 | 12 | 6 | 8 | 8
  Participants with SAEs | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Evaluate Immunogenicity of Multiple Dosage Levels and Dosing Regimens of H56:IC31 - CD4+ ICS (LTBI-negative)
Description: LTBI: Latent TB Infection QFT: QuantiFERON-TB Gold Plus (QFT-Plus) is an in vitro diagnostic aid for detection of Mycobacterium tuberculosis infection Percent Antigen-specific T Cell DMSO-subtracted Cytokine Response Change from Baseline 13-color ICS assay using PBMCs T Cell: CD4+ Stimulation Antigen: Total Cytokine: Any
Time Frame: Day 292
Population: Immunogenicity analysis set: LTBI-negative at baseline
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | 2-Dose Placebo | 2-Dose 5/500 H56/IC31nmol | 2-Dose 15/500 H56/IC31nmol | 2-Dose 50/500 H56/IC31nmol | 3-Dose Placebo | 3-Dose 5/500 H56/IC31nmol
Number analyzed (Participants) | 4 | 13 | 14 | 14 | 3 | 6
Percentage of change from baseline | 0.002 (0.018) | 0.088 (0.104) | 0.027 (0.031) | 0.031 (0.047) | 0.012 (0.014) | 0.045 (0.056)

3. Secondary Outcome: Evaluate Immunogenicity of Multiple Dosage Levels and Dosing Regimens of H56:IC31 - CD4+ ICS (LTBI-positive)
Description: Percent Antigen-specific T Cell DMSO-subtracted Cytokine Response Change from Baseline.
  13-color ICS assay using PBMCs. T Cell: CD4+ Stimulation Antigen: Total Cytokine: Any
Time Frame: Day 292
Population: Immunogenicity analysis set: LTBI-positive at baseline
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | 2-Dose Placebo | 2-Dose 5/500 H56/IC31nmol | 3-Dose Placebo | 3-Dose 5/500 H56/IC31nmol
Number analyzed (Participants) | 4 | 10 | 4 | 8
Percentage of change from baseline | 0.005 (0.020) | 0.068 (0.052) | 0.027 (0.022) | 0.097 (0.170)

4. Secondary Outcome: Evaluate Immunogenicity of Multiple Dosage Levels and Dosing Regimens of H56:IC31 - IFN-gamma ELISpot
Description: DMSO-subtracted Antigen-specific IFN-gamma ELISpot Response (SFU - Background/10^6 PBMC) Change from Baseline LTBI Status at Baseline: Total Stimulation Antigen: Total
Time Frame: Day 292
Population: Immunogenicity analysis set
Measure: Mean (Standard Deviation); unit: Number of spots per well
Arm/Group | 2-Dose Placebo | 2-Dose 5/500 H56/IC31nmol | 2-Dose 15/500 H56/IC31nmol | 2-Dose 50/500 H56/IC31nmol | 3-Dose Placebo | 3-Dose 5/500 H56/IC31nmol
Number analyzed (Participants) | 8 | 21 | 13 | 12 | 7 | 13
Number of spots per well | 82.7 (223.6) | 209.0 (221.8) | 57.9 (162.2) | 110.0 (92.0) | -53.1 (79.8) | 167.4 (364.8)

5. Secondary Outcome: Evaluate Kinetics of QuantiFERON®-TB Gold Test (QFT) Responses in LTBI-negative Participants
Description: QFT results were summarized using subject count (percentage) for qualitative results.
  Number of participants QFT-positive at any time point.
Time Frame: Up to Study Day 292
Population: Conversion of LTBI-negative at baseline to LTBI-positive due to H56:IC31 expression of ESAT-6 (antigen in QFT assay).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QFT Neg | 2-Doses 5/500 QFT Neg | 2-Doses 15/500 | 2-Doses 50/500 | 3-Doses 5/500 QFT Neg
Number analyzed (Participants) | 9 | 15 | 15 | 15 | 12
Participants | 2 | 7 | 6 | 6 | 7

ADVERSE EVENTS:
Time Frame: 10 months
Description: Systematic Assessment - includes diary cards, scheduled visits and lab tests Non-systematic Assessment also collected through self reporting
Groups:
- 2-Dose Placebo: Placebo QFT neg and pos
- 2-Dose 5/500 H56ug/IC31nmol: 2-Dose 5/500 H56ug/IC31nmol, QFT neg and pos
- 2-Dose 15/500 H56ug/IC31nmol: 2-Dose 15/500 H56ug/IC31nmol, QFT negative
- 2-Dose 50/500 H56ug/IC31nmol: 2-Dose 50/500 H56ug/IC31nmol, QFT negative
- 3-Dose Placebo: 3-Dose Placebo QFT neg and pos
- 3-Dose 5/500 H56ug/IC31nmol: 3-Dose 5/500 H56ug/IC31nmol, QFT neg and pos
Arm/Group | 2-Dose Placebo | 2-Dose 5/500 H56ug/IC31nmol | 2-Dose 15/500 H56ug/IC31nmol | 2-Dose 50/500 H56ug/IC31nmol | 3-Dose Placebo | 3-Dose 5/500 H56ug/IC31nmol
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/27 | 0/15 | 0/15 | 0/8 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/27 | 0/15 | 0/15 | 0/8 | 0/24
Other Adverse Events (participants affected / at risk) | 9/9 | 25/27 | 15/15 | 15/15 | 6/8 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-Dose Placebo (N=9) | 2-Dose 5/500 H56ug/IC31nmol (N=27) | 2-Dose 15/500 H56ug/IC31nmol (N=15) | 2-Dose 50/500 H56ug/IC31nmol (N=15) | 3-Dose Placebo (N=8) | 3-Dose 5/500 H56ug/IC31nmol (N=24)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-Dose Placebo (N=9) | 2-Dose 5/500 H56ug/IC31nmol (N=27) | 2-Dose 15/500 H56ug/IC31nmol (N=15) | 2-Dose 50/500 H56ug/IC31nmol (N=15) | 3-Dose Placebo (N=8) | 3-Dose 5/500 H56ug/IC31nmol (N=24)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 5 (5) | 3 (6) | 5 (7) | 2 (3) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 14 (19) | 5 (10) | 8 (11) | 1 (1) | 7 (12)
Injection site swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 2 (3) | 3 (4)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory rate increased (Investigations) | 3 (5) | 13 (25) | 13 (21) | 11 (19) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 5 (6) | 2 (2) | 2 (2) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (7) | 2 (2) | 4 (4) | 1 (1) | 4 (4)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-05-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT01865487/Prot_000.pdf